CLINICAL TRIAL: NCT01982474
Title: Phase I Study of Allergen-Specific Intralymphatic Immunotherapy in the United States
Brief Title: Safety of Lymph Node Injection for Allergen Immunotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amber Patterson (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Amber Patterson, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB13-00409
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — grass pollen extract, alum-adsorbed; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Grass pollen extract injection (Experimental): Grass pollen extract injected intralymphatically q 4 weeks x 3
  Interventions: Biological: Grass pollen extract
- Placebo injection (Placebo Comparator): Normal saline injected intralymphatically q 4 weeks x 3
  Interventions: Other: Placebo injection
- Observational group (No Intervention): Subjects already receiving traditional subcutaneous allergy immunotherapy for grass pollen, being observed for safety of their subcutaneous injections. Not receiving active intervention during this study.

INTERVENTIONS:
Biological: Grass pollen extract — Grass pollen extract injected intralymphatically q 4 weeks x 3
  Arms: Grass pollen extract injection
Other: Placebo injection — Normal saline injected intralymphatically q 4 weeks x 3
  Other Names: Normal saline
  Arms: Placebo injection

SUMMARY:
The purpose of this study is to determine safety of allergy immunotherapy lymph node injections for grass pollen allergies.

DETAILED DESCRIPTION:
Specific immunotherapy (SIT) has been used in the treatment of allergic disease for over one hundred years. SIT for environmental allergies consists of allergen extracts that have been traditionally administered by subcutaneous or sublingual routes to both children and adults. In the United States, subcutaneous immunotherapy (SCIT) is currently the only FDA-approved route of administration for allergenic extracts. In recent years, a novel method of administering allergen immunotherapy, intralymphatic immunotherapy (ILIT), has been developed, which has shown to be safer, more efficacious, and less painful than traditional SCIT. ILIT can dramatically decrease treatment time from 3 - 5 years to 8 weeks. It has only been studied in European adults. The aim of this project is to study efficacy and safety of intralymphatic immunotherapy in adolescents and young adults with allergic rhinoconjunctivitis, using currently available allergen extracts. Patients with clinical history suspicious for rhinitis with or without conjunctivitis, correlating with positive allergy skin and/or blood tests to grass pollen, will be randomized to either placebo (normal saline) or treatment (Center-Al grass pollen extract) arms. A total of 3 injections over eight weeks will be administered intralymphatically. A third arm will include an observational group of grass-allergic subjects already receiving SCIT for 1 year. Primary outcome will be comparison of a safety score between arms 1 and 2. We will follow adverse events, as well as serum markers for Th2 and Th1 phenotypes, and objective respiratory measures (spirometry and FeNO) in those with asthma. Visits will occur at baseline for screening/enrollment, on day 0/week4/week 8 for injections (injection visit for arms 1 and 2 only), and for follow-up at 12 weeks and near end of grass pollen season. A substudy will evaluate participants one-year after completing ILIT injections by obtaining repeat serum biomarker levels and interval change in medical history. Results could help in dramatically decreasing treatment time, as well as increasing safety of allergen immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-24 years
* Bothersome nasal, ocular, and/or respiratory symptoms correlating with grass pollen season (summer)
* Grass pollen allergic (+ skin prick test [wheal ≥ 3 mm larger than negative control] or specific IgE [minimum 0.35 kU/L] to grass pollen [Timothy or a northern pasture grass mix containing Timothy])
* Informed consent obtained and signed
* Informed assent (as appropriate) obtained and signed
* Understanding of study procedures
* Ability to comply with study procedures for the entire length of the study
* For inclusion in observational group (arm 3), must have initiated SCIT containing grass pollen 12 - 18 months prior to grass pollen season 2014 (ex. started SCIT any time Dec 2012 - May 2013). This group was included for comparison between traditional IT and ILIT, and these subjects will continue SCIT during this study. Since patients undergoing SCIT may not see clinical response to therapy until 12 months, we selected this time point to better compare with the more rapid immunologic and clinical changes expected with ILIT.

Exclusion Criteria:

* Significant year-round allergy symptoms and year-round symptoms without worsening during grass pollen season (summer). (Exception: intermittent year-round symptoms with significant worsening during summer is acceptable for inclusion).
* Blood donation or surgery within the previous 30 days of baseline/enrollment, visit #1.
* Use of investigational drugs within the previous 90 days
* Pregnancy or nursing
* Mastocytosis
* Significant cardiovascular, hepatic, renal, autoimmune, hematological, or active infectious disease
* History of malignancy, hypertension, use of immunosuppressive agents, beta-blockers, ACE inhibitors, or tricyclic antidepressants
* Pulmonary disease, including moderate to severe, perennial asthma (FEV1 < 80% predicted) and perennial use of inhaled corticosteroids (exception: seasonal allergic asthma will not be excluded)
* Previous IT (exception: those in observational arm currently on grass SCIT).
* No readily accessible inguinal lymph nodes

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe Adverse Events as a Measure of Safety and Tolerability | Final data regarding adverse events will be assessed one week after the final injection (approximately 3 months after initial injection).

CONTACTS AND LOCATIONS:
Overall Officials: Amber M Patterson, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Background] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Background] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Derived] Patterson AM, Bonny AE, Shiels WE 2nd, Erwin EA. Three-injection intralymphatic immunotherapy in adolescents and young adults with grass pollen rhinoconjunctivitis. Ann Allergy Asthma Immunol. 2016 Feb;116(2):168-70. doi: 10.1016/j.anai.2015.11.010. Epub 2015 Dec 17. No abstract available. PMID 26706294